CLINICAL TRIAL: NCT06733935
Title: A Phase 1/2 Study of NKX019, a CD19 Chimeric Antigen Receptor Natural Killer (CAR NK) Cell Therapy, in Subjects With Immune-Mediated Diseases
Brief Title: A Phase 1/2 Study of NKX019 in Subjects With Immune-Mediated Diseases (Ntrust-2)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nkarta, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ntrust-2
Record Dates: First submitted 2024-12-04; First posted 2024-12-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Antineutrophil Cytoplasmic Antibody-Associated Vasculitis
Keywords: CD19; CAR; Allogeneic; NKX019; Natural Killer Cells; Interleukin-15; IL-15; Cell Therapy; Immunotherapy; Adoptive cell therapy; Scleroderma; Myositis; AAV; Systemic Sclerosis; Idiopathic Inflammatory Myopathies; Antineutrophil Cytoplasmic Antibody (ANCA)-Associated Vasculitis; Ntrust-2
MeSH Terms: conditions — Scleroderma, Systemic; Myositis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Scleroderma, Diffuse | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKX019 - CAR NK cell therapy (Experimental): Phase 1/2: NKX019 plus fludarabine and cyclophosphamide
  Interventions: Drug: NKX019; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: NKX019 — NKX019 is an investigational allogeneic CD19-Directed CAR NK
Drug: Fludarabine — Lymphodepletion
Drug: Cyclophosphamide — Lymphodepletion

SUMMARY:
This is a Phase 1/2, open-label, multi-center, multi-cohort, non-randomized dose escalation and dose expansion basket study to determine the safety and tolerability of NKX019 (allogeneic CAR NK cells targeting CD19) in participants with autoimmune diseases.

DETAILED DESCRIPTION:
Dose escalation of NKX019 will utilize a "3+3" design to determine the recommended dose(s) for expansion for enrolling additional participants across indications. The study will evaluate safety and tolerability, preliminary efficacy, pharmacokinetics, pharmacodynamics, and immunogenicity in participants with autoimmune diseases. Participants will receive a cycle consisting of lymphodepletion with fludarabine and cyclophosphamide (Flu/Cy) followed by three doses of NKX019. Participants who are cytopenic may receive a modified lymphodepletion regimen of Cy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤70
2. For participants taking corticosteroids, the prednisone (or equivalent) dose must be ≤40 mg/day at 6 weeks prior to Screening and stable for ≥ 14 days before start of Screening
3. For subjects on immunosuppressives or immunomodulators (other than corticosteroids), all doses must be stable for ≥ 4 weeks prior to Screening

SSc:

1. Meets the 2013 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology (EULAR) classification criteria for SSc
2. Meet criteria a and/or b:

   1. Severe skin involvement defined as mRSS ≥ 30 or active skin disease defined as mRSS ≥ 15 at screening and one or more of the following within the prior 6 months of screening:

      * An increase in mRSS of ≥ 3 units
      * Involvement of 1 new body area with ≥ 2 mRSS units
      * 2 new body areas with ≥ 1 mRSS unit
   2. Moderate to severe Interstitial Lung Disease (ILD) defined by evidence of ILD on High-resolution computed tomography (HRCT) and FVC < 70% of predicted or DLCO (hemoglobin or alveolar volume corrected) < 70% of predicted or ILD on HRCT and progressive ILD meeting at least 2 of the following 3 criteria within the prior 6 months of screening:

      * Worsening respiratory symptoms
      * Evidence of progression on HRCT, or
      * Evidence of absolute decline in FVC ≥ 5% (Raghu et al 2022)
3. Presence of anti-nuclear antibody ≥ 2 x upper limit of normal (ULN)
4. 10 years or less since the first non-Raynaud's sign or symptom
5. Inadequate response or intolerance to at least one treatment, including cyclophosphamide, methotrexate, MMF/mycophenolic acid, nintedanib, rituximab, or tocilizumab

IIM:

1. Diagnosis for IIM as per 2017 ACR/EULAR Classification Criteria
2. One positive myositis antibody
3. Activity defined as manual muscle testing (MMT-8) score <136/150
4. Creatinine kinase or aldolase ≥ 1.5 x ULN and Clinician Global Assessment ≥ 2 cm with at least one of the following:

   1. Evidence on magnetic resonance imaging (MRI) of active myositis within the last 6 months
   2. Electromyography (EMG) with active myositis within the last 6 months
   3. Muscle Biopsy of active myositis within last 6 months
5. Refractory disease defined as ≥ 6 months failure (or intolerance) to at least 2 immunosuppressive therapies (including glucocorticoids)

AAV:

1. Meets the 2022 ACR/EULAR classification criteria for Granulomatosis with Polyangiitis (GPA) (Robson 2022) or Microscopic Polyangiitis (MPA) (Suppiah 2022)
2. Relapsed or refractory AAV despite repeated treatment with immunosuppressive agents or requiring prolonged and/or repeated courses of unacceptable doses of glucocorticoids to maintain disease control
3. Positive test for anti-proteinase-3 (PR3-ANCA) or anti-myeloperoxidase (MPO-ANCA) at screening
4. Have at least one "major" item, or at least 3 other items, or at least 2 renal items on the BVAS version 3

Exclusion Criteria:

1. eGFR < 45 ml/min/1.73m2
2. Currently requiring renal dialysis or expected to require dialysis during the study period
3. Previous solid organ or hematopoietic cell transplant or planned transplant within study treatment period
4. Congenital or acquired immunodeficiency resulting in severe infection or those receiving chronic immunoglobulin replacement therapy
5. Liver disease or dysfunction, including cirrhosis and/or bilirubin ≥ 3 times the upper limit of normal
6. Pulmonary comorbidity including chronic obstructive pulmonary disease or asthma requiring daily oral steroids, resting hypoxemia (<92% oxygen saturation via pulse oximetry) on room air, or significant smoking history (i.e. >10 pack/year) with active pulmonary disease
7. Patients with ILD with any of the following:

   1. Requires supplemental oxygen therapy
   2. FVC <=45% of predicted
   3. Diffusing capacity of the lung (DLCO) corrected for alveolar volume (AV) ≤ 40% of predicted at screening (per Investigator or Sponsor judgement)
8. White blood cell count < 3,000/mm^3; hemoglobin levels ≤ 9 g/dL; absolute neutrophil count (ANC) ≤ 2,000/mm^3; platelet count ≤ 100,000/mm^3, and blood transfusion within 60 days prior to LD
9. Major cardiac disease, abnormalities, or interventions as defined by, but not limited to:

   1. Uncontrolled angina or unstable life-threatening arrhythmias
   2. History of myocardial infarction within 12 weeks prior to the first dose of NKX019
   3. Any prior coronary artery bypass graft surgery
   4. ≥ Class III New York Heart Association (NYHA) congestive heart failure (CHF), significantly decreased ejection fraction (EF ≤ 40%), or severe cardiac insufficiency
   5. Prolongation of the QT interval corrected for heart rate (QTc) (Fridericia) interval of > 480 msec
   6. Peripheral artery bypass graft surgery, pulmonary embolism, or other ≥ Grade 2 thrombotic or embolic events within 12 weeks prior to the first dose of NKX019
10. Active bleeding disorders
11. Any overlapping autoimmune condition for which the condition or the treatment of the condition may affect the study assessments or outcomes (eg, anti-GBM antibody glomerulonephritis or any condition for additional immunosuppression is indicated); clinically significant conditions that could cause a secondary nephropathy (eg, infections, liver disease, tumors or drugs); or kidney biopsy-confirmed significant renal disease other than disease under study (eg, diabetic nephropathy, hypertensive nephropathy). Overlapping conditions for which the condition or treatment is not expected to affect assessments or outcomes (eg, Sjögren's syndrome, rheumatoid arthritis) are not excluded
12. Pregnancy, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions
13. Current infection requiring active systemic anti-infective therapy or recent acute infection requiring systemic therapy within 30 days of planned LD
14. History of positive HIV test at screening, Hepatitis B or C positive at screening, active tuberculosis (TB) or latent TB requiring suppressive therapy
15. Major surgery within 28 days prior to the first dose of NKX019
16. Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia but have been treated with conization or loop electrosurgical excision procedure and have had a normal repeat Papanicolaou test are allowed
17. Prior cellular therapy
18. Central nervous system (CNS) comorbidity or any autoimmune disease with CNS involvement within 90 days prior to the first dose of NKX019 as well as evidence of CNS related autoimmune manifestations within 1 year prior to screening
19. Immunosuppressive / immunomodulatory therapies for disease under study within 14 days or 5 half-lives of the drug (whichever is shorter), prior to LD, with notable exceptions a. For those participants on B-cell-depleting or B-cell-modulating drugs (eg, rituximab, belimumab), the participants must have received first dose ≥6 months prior to LD

SSc Exclusion Criteria:

1. Moderate-to-severe Pulmonary arterial hypertension (PAH) on right heart catheterization requiring PAH specific treatment. Those participants with mild PAH (as defined by the 2022 ECS/ERS Guidelines, [Humbert 2023]) well controlled on therapy can be enrolled
2. Gastrointestinal (GI) dysmotility requiring total parenteral nutrition (TPN)
3. Anti-centromere Ab positive
4. Renal crisis or Pericardial tamponade within 6 months prior to enrollment
5. Current gangrene of a digit

IIM Exclusion Criteria:

1. Severe proximal muscle atrophy of upper or lower extremity on Magnetic Resonance Imaging (MRI) or clinical exam
2. MMT-8 of ≤ 80
3. Findings of muscular inflammation or myopathy due to another cause, such as inclusion body myositis, cancer-associated myositis (myositis diagnosed within 2 years of cancer), amyloid myopathy, muscular dystrophy, metabolic myopathies, or myositis in the context of significant overlap with another systemic IIM rheumatologic disease (overlap myositis), except with Sjögren's syndrome
4. Generalized severe musculoskeletal or neuro-muscular conditions other than IIM

AAV Exclusion Criteria:

1. Alveolar hemorrhage requiring invasive pulmonary ventilation support
2. Required dialysis or plasma exchange within 12 weeks prior to screening
3. Any other known disease that may interfere with the assessments including eosinophilic GPA (Churg-Strauss), anti-glomerular basement membrane, systemic lupus erythematosus, IgA vasculitis (Henoch Schönlein), rheumatoid vasculitis, or cryoglobulinemic vasculitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicities (DLTs) [Safety and Tolerability] | The first 28 days after the first NKX019 dose
  Incidence of DLTs will be evaluated
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the first administration of NKX019 until the last administration of any study treatment + 30 days
  Incidence and severity of treatment-emergent adverse events will be evaluated

SECONDARY OUTCOMES:
For all participants with Interstitial Lung Disease (ILD) | Up to 2 years after NKX019 infusion
  Change from baseline in % predicted forced vital capacity (FVC) over time
For all participants with Interstitial Lung Disease (ILD) | Up to 2 years after NKX019 infusion
  Change from baseline % predicted CO (DLCO) corrected for alveolar volume (AV) over time
For all participants with Interstitial Lung Disease (ILD) | Up to 2 years after NKX019 infusion
  Time to and proportion of participants with improvement in FVC by ≥10%
For all participants with Interstitial Lung Disease (ILD) | Up to 2 years after NKX019 infusion
  Time to and proportion of participants with ILD progression
For all participants with Systemic Sclerosis (SSc) | Up to 2 years after NKX019 infusion
  Change from baseline in modified Rodnan skin score (mRSS)
For all participants with Systemic Sclerosis (SSc) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving revised Composite Response Index (rCRISS) 25, 50 and 70 at 3, 6, and 12 months compared to baseline
For all participants with Systemic Sclerosis (SSc) | Up to 2 years after NKX019 infusion
  Change from baseline modified EULAR (European Alliance of Associations for Rheumatology) Scleroderma
For all participants with Systemic Sclerosis (SSc) | Up to 2 years after NKX019 infusion
  Trials and Research Activity Index (EUSTAR AI) over time
For all participants with Systemic Sclerosis (SSc) | Up to 2 years after NKX019 infusion
  Change from baseline University of California Los Angeles Gastrointestinal Tract (UCLA GIT) 2.0 assessments over time
For all participants with Idiopathic Inflammatory Myopathies (IIM) | Up to 2 years after NKX019 infusion
  Change from baseline in manual muscle testing (MMT) over time
For all participants with Idiopathic Inflammatory Myopathies (IIM) | Up to 2 years after NKX019 infusion
  Change from baseline and normalization of muscle enzymes over time
For all participants with Idiopathic Inflammatory Myopathies (IIM) | Up to 2 years after NKX019 infusion
  Change from baseline Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) score (dermatomyositis only) over time
For all participants with Idiopathic Inflammatory Myopathies (IIM) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving a mild, moderate, or major (20, 40, 60 points) clinical response by Total Improvement Score (TIS) at 3, 6, and 12 months (including assessment of change from baseline in TIS components)
For all participants with ANCA-Associated Vasculitis (AAV) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving Birmingham Vasculitis Activity Score (BVAS) remission at 3, 6, and 12 months
For all participants with ANCA-Associated Vasculitis (AAV) | Up to 2 years after NKX019 infusion
  Change from baseline BVAS over time
For all participants with ANCA-Associated Vasculitis (AAV) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving clinical remission Off Therapy (CROffT) at 3, 6, and 12 months
For all participants with ANCA-Associated Vasculitis (AAV) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving clinical remission On Therapy (CROnT) at 3, 6, and 12 months
For all participants with ANCA-Associated Vasculitis (AAV) | Up to 2 years after NKX019 infusion
  Proportion of participants achieving low disease activity state (LDAS) at 3, 6, and 12 months (Delvino 2023), change from baseline ESR, CRP over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of participants requiring rescue therapy (all participants) over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of participants who are steroid free (IIM, AAV) over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Cumulative corticosteroid dose (IIM, AAV) over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of participants receiving 5 mg daily prednisone (or equivalent) over time
Evaluation of the effect of treatment on background therapies | Up to 2 years after NKX019 infusion
  Proportion of participants receiving 7.5 mg daily prednisone (or equivalent) over time
Pharmacokinetics parameter: maximum concentration (Cmax) | Up to 2 years after NKX019 infusion
Pharmacokinetics parameter: Time-to-maximum concentration (Tmax) | Up to 2 years after NKX019 infusion
Pharmacokinetics parameter: Area under the curve (AUC) | Up to 2 years after NKX019 infusion
Pharmacokinetics parameter: Half-life (t1/2) | Up to 2 years after NKX019 infusion
Duration of persistence of NKX019 in peripheral blood | Up to 2 years after NKX019 infusion
Assess humoral immunogenicity over time with validated methods that include: a cell-based flow cytometry assay for anti-NKX019 antibodies and an antigen bead-assay using flow cytometry for detection of anti-HLA antibodies | Up to 2 years after NKX019 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nkarta Study Director, Study Director — Nkarta, Inc.
Locations (12):
- United States (11):
  - Nkarta Investigational Site, Orange, California
  - Nkarta Investigational Site, Miami, Florida
  - Nkarta Investigational Site, Plantation, Florida
  - Nkarta Investigational Site, Chicago, Illinois
  - Nkarta Investigational Site, Fairway, Kansas
  - Nkarta Investigational Site, Ann Arbor, Michigan
  - Nkarta Investigational Site, Minneapolis, Minnesota
  - Nkarta Investigational Site, Hackensack, New Jersey
  - Nkarta Investigational Site, Stony Brook, New York
  - Nkarta Investigational Site, Dallas, Texas
  - Nkarta Investigational Site, Houston, Texas
- Nkarta Investigational Site, Manatí, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Ntrust-2 Study for Autoimmune Diseases — https://www.ntrust2.com/